CLINICAL TRIAL: NCT02356874
Title: Exercise for SpondyloArthritis (SpA) - the ESpA Study The Effect of a Supervised Exercise Intervention on Disease Activity and Cardiovascular Risk in Patients With SpA - A Multicenter Randomized Controlled Trial
Brief Title: The Effect of Exercise on Disease Activity and Cardiovascular Risk for Patients With Axial SpondyloArthritis
Acronym: ESpA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: University of Oslo (Other); Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Silje H Sveaas, PT, PhD, PhD, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 97026: The ESpA study
Record Dates: First submitted 2015-01-21; First posted 2015-02-05 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2017-02

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Exercise group (Experimental): Exercise
  Interventions: Behavioral: Exercise
- Control group (No Intervention): Participants in the control group will be asked to continue their usual physical activity habits

INTERVENTIONS:
Behavioral: Exercise — An exercise program for 40-60 minutes three times a week in 3 months. Twice a week the exercise sessions will be supervised by a physiotherapist and these sessions will consist of endurance and strength training. The endurance training will be high intensity interval training on a treadmill. And strength training with external load for the major muscle groups (individually adapted: six exercises, eight to ten repetitions maximum, two to three sets). Once a week the participants will exercise individually for a minimum of 40 minutes of endurance exercise.
  Arms: Exercise group

SUMMARY:
The overall aim of this multicenter randomised controlled trial (RCT) is to investigate if exercise can modify the disease course and prevent comorbidity in patient with spondyloarthritis (SpA).

DETAILED DESCRIPTION:
International guidelines recommend exercise as a cornerstone in the management of SpA. Due to the typical features of SpA with reduced spinal mobility, the main focus for exercise has been flexibility exercise. Exercise trials for this patient group have mainly aimed at improving spinal mobility and there is limited evidence of the potential effects of exercise on disease pathogenesis and CVD risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of axial SpA (the Assessment of SpondyloArthritis International Society classification criteria) confirmed by a rheumatologist
2. Age, 18-70 -years
3. Steady medication for ≥3 months
4. Moderate disease activity defined as a BASDAI score of ≥3.5 or a patient global score ≥3.5
5. Not participated in a structured endurance and strength exercise program during the last 6 months (>1 hour/week)

Exclusion Criteria:

1. Severe co-morbidity which involves reduced exercise capacity and/or contraindications for physical activity as per American College of Sports Medicine guidelines for exercise testing
2. Not able to participate in weekly exercises sessions
3. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Disease activity | 3 months
  The Ankylosing Spondylitis Disease Activity Score (ASDAS) and the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)

SECONDARY OUTCOMES:
Blood samples | 3 months (all analyses) 12 months (only CRP and ESR)
  General and specific markers of inflammation and cardiovascular risk
Spinal mobility | 3 months
  The Bath Ankylosing Spondylitis Metrology Index (BASMI). BASMI includes five measurements of flexibility in the spine, neck and hips.
Physical function | 3 months and 12 months
  The Bath Ankylosing Spondylitis functional Index (BASFI).
Cardiorespiratory fitness | 3 months
  Maximal walking test on a treadmill for estimation of maximal oxygen uptake.
Body composition | 3 months
  Body weight, body height, waist and hip circumference. DXA scan of a sample of patients.
Arterial stiffness | 3 months
  Pulse wave velocity and argumentation Index
Endothelial function | 3 months
  Digital plethysmography using the non-invasive ADMAR apparatus (sample of participants)
Blood pressure | 3 months
General health | 3 months and 12 months
  Assessed with the general health questionnaire (GHQ-12)
Health related quality of life | 3 months and 12 months
  Euro Quol 5D (EQ5D)
Physical activity level | 3 months and 12 months
  Questionaire of frequency, intensity and duration of physical activity
Self-efficacy for physical activity | 3 months and 12 months
  Questionnaire
Fatigue | 3 months and 12 months
  The fatigue severity scale and the SF-36 vitality scale (version 1)
Sleep | 3 months and 12 months
  Pittsburgh Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Hanne H Dagfinrud, PhD, Principal Investigator — Nationonal Advisory Unit on Rehabilitation in Rheumatology, Departement of Rheumatology, Diakonhjemmet Hospital
Locations (4):
- Norway (3):
  - Martina Hansens Hospital AS, Bærum
  - Diakonhjemmet Hospital AS, Oslo
  - University Hospital of North Norway, Tromsø
- University of Gotenburg, Gothenburg, Sweden

REFERENCES:
- [Derived] Fongen C, Dagfinrud H, Bilberg A, Sveaas SH. Reduced sleep quality is highly prevalent and associated with physical function and cardiorespiratory fitness in patients with axial spondyloarthritis: a cross-sectional study. Scand J Rheumatol. 2024 Mar;53(2):130-139. doi: 10.1080/03009742.2023.2281069. Epub 2023 Dec 14. PMID 38095452
- [Derived] Bilberg A, Dagfinrud H, Sveaas SH. Supervised Intensive Exercise for Strengthening Exercise Health Beliefs in Patients With Axial Spondyloarthritis: A Multicenter Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2022 Jul;74(7):1196-1204. doi: 10.1002/acr.24556. Epub 2022 Apr 17. PMID 33423392
- [Derived] Sveaas SH, Dagfinrud H, Berg IJ, Provan SA, Johansen MW, Pedersen E, Bilberg A. High-Intensity Exercise Improves Fatigue, Sleep, and Mood in Patients With Axial Spondyloarthritis: Secondary Analysis of a Randomized Controlled Trial. Phys Ther. 2020 Aug 12;100(8):1323-1332. doi: 10.1093/ptj/pzaa086. PMID 32367124
- [Derived] Fongen C, Dagfinrud H, Bilberg A, Pedersen E, Johansen MW, van Weely S, Hagen KB, Sveaas SH. Responsiveness and Interpretability of 2 Measures of Physical Function in Patients With Spondyloarthritis. Phys Ther. 2020 Apr 17;100(4):728-738. doi: 10.1093/ptj/pzaa004. PMID 31944251
- [Derived] Sveaas SH, Dagfinrud H, Johansen MW, Pedersen E, Wold OM, Bilberg A. Longterm Effect on Leisure Time Physical Activity Level in Individuals with Axial Spondyloarthritis: Secondary Analysis of a Randomized Controlled Trial. J Rheumatol. 2020 Aug 1;47(8):1189-1197. doi: 10.3899/jrheum.190317. Epub 2019 Nov 15. PMID 31732552
- [Derived] Sveaas SH, Bilberg A, Berg IJ, Provan SA, Rollefstad S, Semb AG, Hagen KB, Johansen MW, Pedersen E, Dagfinrud H. High intensity exercise for 3 months reduces disease activity in axial spondyloarthritis (axSpA): a multicentre randomised trial of 100 patients. Br J Sports Med. 2020 Mar;54(5):292-297. doi: 10.1136/bjsports-2018-099943. Epub 2019 Feb 11. PMID 30745314